CLINICAL TRIAL: NCT06609213
Title: Oral Intake of Enteral Nutrition Formula Preceding Placement and Feeding Via G-Tube and Its Impact on Formula Intolerance in pALS
Brief Title: Oral Intake of Enteral Nutrition Formula Preceding Placement and Feeding Via GTube and Its Impact on Formula Intolerance in pALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrea Charvet (Other)
Collaborators: Nova Southeastern University (Other)
Responsible Party: Sponsor-Investigator, Andrea Charvet, Assistant Professor, Nova Southeastern University
Organization: Nova Southeastern University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-464-NSU; 334957 (Other Grant/Funding Number: Nova Southeastern University)
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Amyotrophic Lateral Sclerosis; Gastrointestinal Intolerance; Enteral Nutrition Therapy
Keywords: amyotrophic lateral sclerosis; ALS; Gtube; enteral nutrition; feeding intolerance; EN intolerance; enteral nutrition intolerance; gastrointestinal symptoms; percutaneous endoscopic gastrostomy; PEG
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: This single arm intervention study will utilize validated indicators combined with clinical expertise to assess GI symptoms of feeding intolerance before and after the intervention in a way that each patient serves as their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): This is a single arm study in which all participants receive the intervention.
  Interventions: Other: Medical Food

INTERVENTIONS:
Other: Medical Food — Enteral nutrition formula will be used both by mouth and via feeding tube. This product is considered a medical food.

SUMMARY:
The main objective of the proposed study is to evaluate if oral intake of EN formula preceding Gtube placement will impact tolerance upon placement and feeding via Gtube in pALS. This single arm intervention study all participants will receive the intervention and researchers will utilize validated indicators combined with clinical expertise to assess gastrointestinal symptoms of feeding intolerance before and after the intervention.

The main questions this study aims to answer are:

1. Wil participants meeting a greater percentage of their estimated nutritional needs at baseline present a slower disease progression rate and a lower incidence of GI symptoms of feeding intolerance when feeding via Gtube?
2. Will there be significant change in feeding intolerance when oral intake of enteral nutrition formula precedes feeding via Gtube?

This proposed study consists of three stages, as follows:

1. Pre-Intervention: The lead in period of one-week preceding intervention phase I will be timed to initiate 3 weeks before the scheduled Gtube placement procedure. Patients will be advised to maintain their usual food and beverage intake. Dietary intake and GI symptoms data will be collected by research personnel.
2. Phase I: Dietary intake data collected from the pre-intervention stage will be averaged and used to determine the number of cartons of enteral nutrition formula needed to meet the participants estimated nutritional needs. For two weeks +- 2 days participants will be directed to drink the number of cartons of a pre-selected enteral nutrition formula to meet their estimated nutritional needs when combined to their current oral dietary intake. A plant based EN formula (Kate Farms 1.4 Standard) commonly prescribed for pALS was selected to be provided to all patients in the study to keep this variable constant. Weekly data collection of dietary intake and GI symptoms will be ongoing.
3. Phase II: At the end of phase I, patients will undergo a Gtube placement at their selected medical facility. For the following two weeks +- 2 days participants will be directed to feed via Gtube the same number of cartons of the enteral nutrition formula used orally on phase I and make no changes to their current oral intake.

DETAILED DESCRIPTION:
Brief Background:

Amyotrophic lateral sclerosis (ALS) is a progressive and fatal neurodegenerative disease. Over 82% of patients with ALS (pALS), develop dysphagia as disease progresses. Dysphagia leads to a decrease in oral intake associated with the fear of choking and long duration of meals, which results in weight loss and consequently malnutrition. Malnutrition is associated with a shorter survival time in pALS. Feeding via a gastrostomy tube (Gtube) bypasses oral intake and helps individuals maintain adequate nutrition. Research shows that Gtube usage significantly increases survival time in pALS. Despite a low risk for major complications with a Gtube placement, enteral nutrition (EN) intolerance is reported in 27-38% of hospitalized and critically ill patients. Intolerance, frequently defined by the presence of gastrointestinal (GI) symptoms, contributes to poor adherence with nutritional recommendations, further weight loss and greater risk of malnutrition. Currently, there is no data of the prevalence of EN intolerance among pALS or evidence on the impact of oral intake of EN formula on intolerance. Data from the Cathy J. Husman ALS Center at NSU Health show that 28.6% of the patients who had a Gtube tube placed changed EN formula due to intolerance.

Objectives:

The primary aim of this single-arm study is to evaluate whether oral intake of EN formula preceding Gtube placement will impact tolerance upon placement and feeding via Gtube in pALS. GI symptoms and dietary intake will be assessed before and after the intervention in a proposed sample of 22 pALS. This study involves a multidisciplinary collaboration of professionals in our clinic. It was designed with the teams expertise and includes pertinent indicators to assess EN intolerance in a population with great needs and insufficient research. Potential therapeutic strategies learned from this study can be incorporated into clinical practice guidelines much needed in the management of Gtube usage to minimize malnutrition, increase survival time, and improve quality of life in pALS.

Specific Aims:

Aim 1: Analyze dietary intake before and after placement and feeding via Gtube and determine its relationship with disease progression and GI symptoms of feeding intolerance.

Aim 2: Evaluate GI symptoms of feeding intolerance at baseline, during oral intake of EN formula, and after placement and feeding via Gtube.

Study Design:

In this single arm intervention study participants will be recruited during their routine multidisciplinary visit at the NSU Health ALS Center. The intervention will take place as part of the daily feeding routine of the patients, at their desired location. This proposed study consists of three stages: pre-intervention, phase I, and phase II. Assessments will be completed by the patients and/or their caregivers at home and collected weekly by research personnel via phone calls and email. The primary outcome measure will be gastrointestinal symptoms of EN intolerance. Secondary outcome measures include dietary intake, body mass index (BMI), and ALS Functional Rating Scale (ALSFRS-R). Treatment fidelity will be assessed at the end of the study.

Experimental Procedures and Outcome Measures

This proposed study consists of three stages, as follows:

1. Pre-Intervention: The lead in period of one-week preceding intervention phase I will be timed to initiate 3 weeks before the scheduled Gtube placement procedure. Patients will be advised to maintain their usual food and beverage intake. Dietary intake and GI symptoms data will be collected as described below.
2. Phase I: Dietary intake data collected from the pre-intervention stage will be averaged and used to determine the number of cartons of enteral nutrition formula needed to meet the participants estimated nutritional needs. For two weeks +- 2 days participants will be directed to drink the number of cartons of a pre-selected enteral nutrition formula to meet their estimated nutritional needs when combined to their current oral dietary intake. Nutritional needs will be estimated using the predictive equation researched and developed by Kasarskis and colleagues to estimate energy requirements of ALS patients. A plant based EN formula (Kate Farms 1.4 Standard) commonly prescribed for pALS was selected to be provided to all patients in the study to keep this variable constant. Weekly data collection of dietary intake and GI symptoms will be ongoing as described below.
3. Phase II: At the end of phase I, patients will undergo a Gtube placement at their selected medical facility. For the following two weeks +- 2 days participants will be directed to feed via Gtube the same number of cartons of the enteral nutrition formula used orally on phase I and make no changes to their current oral intake. Weekly data collection of dietary intake and GI symptoms will be ongoing as described below.

Demographics:

At baseline, the following demographic and clinical information will be obtained: age, biological sex, race, ethnicity, ALS disease onset type and duration (months), height, weight, body mass index (BMI), malnutrition risk (change in BMI from first appointment to current), overall disease severity as indexed by the validated the ALS Functional Rating Scale (ALSFRS) score, and disease progression rate (change in ALSFRS from first appointment to current).

Dietary Intake:

To determine dietary intake of each participant, a food diary will be completed by the participant, with or without the aid of a caregiver, for the duration of the study. Patients and caregivers will be provided instructions on how to complete the food diary and will be directed to record intake at the time of consumption. For each week, the food diary must be completed for a minimum of 3 days and a maximum of 7 days. The weekly intake of selected nutrients will be averaged. A diet analysis software will be utilized to analyze the dietary intake information obtained. Nutritionist Pro, by Axxya Systems, is a software application for nutrition technology and data that uses the Nutrition Raw Database of Foods and Beverages to calculate nutrition values, a system compliant with USA requirements.

Gastrointestinal Symptoms:

Gastrointestinal symptoms of feeding intolerance will be monitored weekly using a clinician-administered survey. The Gastrointestinal Symptom Rating Scale (GSRS) is a 15-item scale that combines each item into five symptom clusters including reflux, abdominal pain, indigestion, diarrhea, and constipation. Patients rate each item on a 7-point Likert scale (from no discomfort at all to very severe discomfort). The recall period is seven days, and it is estimated to take about 3 to 5 minutes to complete. The clinical team will also be monitoring study participants for any significant gastrointestinal event that requires medical attention at any point in time during the study. These will be recorded when the patient contacts the clinic for medical attention, or patient-reported if medical attention is sought elsewhere.

Data Analysis Descriptive statistics will be used to explore dietary intake and the prevalence of GI symptoms of feeding intolerance in pALS. Dietary intake and prevalence of GI symptoms of feeding intolerance before and after placement and feeding via Gtube will be compared within subjects using paired t-test. To assess the relationships between the percentage of estimated nutritional needs met at baseline and disease progression indicators, as well as the incidence of GI symptoms of feeding intolerance after placement and feeding via Gtube, Pearson's correlation will be used (Aim 1). To determine the change in GI symptoms of feeding intolerance at baseline, during oral intake of enteral nutrition formula, and after placement and feeding via Gtube, a one-way repeated measures analysis of variance (ANOVA) will be conducted (Aim2). Statistical analysis will be conducted using SPSS (SPSS Statistics V29, IBM) with statistical significance at p-value less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of possible, probable, or definite ALS or motor neuron disease by the treating neurologist (El-Escorial Revisited).
* Planned tube feeding placement within the following 4 to 6 weeks.

Exclusion Criteria:

* History of Crohns disease, inflammatory bowel disease, irritable bowel syndrome, celiac disease, food allergies and/or sensitivities to any of the formula ingredients, neurodegenerative disease diagnosis outside of ALS, or other concomitant disorder that might contribute to GI symptoms.
* Diagnosis of frontotemporal dementia.
* Nil per oral status.
* Any reason causing the immediate need for a feeding tube placement, including but not limited to severe malnutrition diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal Symptoms | 5 weeks
  Gastrointestinal symptoms of feeding intolerance will be monitored weekly using a clinician-administered survey in-person or via phone interview. The Gastrointestinal Symptom Rating Scale (GSRS) is a 15-item scale that combines each item into five symptom clusters including reflux, abdominal pain, indigestion, diarrhea, and constipation (Svedlund et al., 1988). Patients rate each item on a 7-point Likert scale (from no discomfort at all to very severe discomfort).

SECONDARY OUTCOMES:
Dietary Intake | 5 weeks
  To determine dietary intake of each participant, a food diary will be completed by the participant, with or without the aid of a caregiver, for the duration of the study. Patients and caregivers will be provided instructions on how to complete the food diary and will be directed to record intake at the time of consumption. For each week, the food diary must be completed for a minimum of 3 days and a maximum of 7 days. The weekly intake of selected nutrients will be averaged. A diet analysis software will be utilized to analyze the dietary intake information obtained. Nutritionist Pro, by Axxya Systems, is a software application for nutrition technology and data that uses the Nutrition Raw Database of Foods and Beverages to calculate nutrition values, a system compliant with USA requirements.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Southeastern University, Cathy J, Husman ALS Center, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No
The study protocol does not include a plan to share IPD.

REFERENCES:
- [Background] Li J, Wang L, Zhang H, Zou T, Kang Y, He W, Xu Y, Yin W. Different definitions of feeding intolerance and their associations with outcomes of critically ill adults receiving enteral nutrition: a systematic review and meta-analysis. J Intensive Care. 2023 Jul 5;11(1):29. doi: 10.1186/s40560-023-00674-3. PMID 37408020
- [Background] Marin B, Desport JC, Kajeu P, Jesus P, Nicolaud B, Nicol M, Preux PM, Couratier P. Alteration of nutritional status at diagnosis is a prognostic factor for survival of amyotrophic lateral sclerosis patients. J Neurol Neurosurg Psychiatry. 2011 Jun;82(6):628-34. doi: 10.1136/jnnp.2010.211474. Epub 2010 Nov 19. PMID 21097551
- [Background] Svedlund J, Sjodin I, Dotevall G. GSRS--a clinical rating scale for gastrointestinal symptoms in patients with irritable bowel syndrome and peptic ulcer disease. Dig Dis Sci. 1988 Feb;33(2):129-34. doi: 10.1007/BF01535722. PMID 3123181
- [Background] Jenkins B, Calder PC, Marino LV. A systematic review of the definitions and prevalence of feeding intolerance in critically ill adults. Clin Nutr ESPEN. 2022 Jun;49:92-102. doi: 10.1016/j.clnesp.2022.04.014. Epub 2022 Apr 20. PMID 35623881
- [Background] Gungabissoon U, Hacquoil K, Bains C, Irizarry M, Dukes G, Williamson R, Deane AM, Heyland DK. Prevalence, risk factors, clinical consequences, and treatment of enteral feed intolerance during critical illness. JPEN J Parenter Enteral Nutr. 2015 May;39(4):441-8. doi: 10.1177/0148607114526450. Epub 2014 Mar 17. PMID 24637246
- [Background] Bond L, Ganguly P, Khamankar N, Mallet N, Bowen G, Green B, Mitchell CS. A Comprehensive Examination of Percutaneous Endoscopic Gastrostomy and Its Association with Amyotrophic Lateral Sclerosis Patient Outcomes. Brain Sci. 2019 Sep 4;9(9):223. doi: 10.3390/brainsci9090223. PMID 31487846
- [Background] Blaser AR, Starkopf J, Kirsimagi U, Deane AM. Definition, prevalence, and outcome of feeding intolerance in intensive care: a systematic review and meta-analysis. Acta Anaesthesiol Scand. 2014 Sep;58(8):914-22. doi: 10.1111/aas.12302. Epub 2014 Mar 11. PMID 24611520